CLINICAL TRIAL: NCT00774631
Title: Mild Induced Hypothermia to Treat Severe Community Acquired Meningitis in Adults Admitted to Intensive Care Unit
Brief Title: IHPOTOTAM : Induced HyPOthermia TO Treat Adult Meningitis
Acronym: IHPOTOTAM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor stoppes the study for the security problem.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 060217; AOM 06 038 (Other: French Ministry)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-07

CONDITIONS: Bacterial Meningitis
Keywords: Meningitis; Hypothermia; Intensive care
MeSH Terms: conditions — Meningitis, Bacterial; Meningitis; Hypothermia | interventions — Hypothermia, Induced; Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypothermia (Experimental): mild induced hypothermia (32-34°C) during 48 hours followed by passive rewarming
  Interventions: Procedure: Mild induced hypothermia (32-34°C)
- No hypothermia (Active Comparator): no hypothermia, according to local recommendations and guidelines of medical societies and literature
  Interventions: Procedure: local recommendations and guidelines

INTERVENTIONS:
Procedure: Mild induced hypothermia (32-34°C) — Mild Induced hypothermia:
  Investigators are advised to use the cooling techniques as used in patients with cardiac arrest. Thus, the choice of cooling method will be left to investigators. Hypothermia will be induced by cold saline infusion as described in appendix 5 [6, 48]. Core temperature will be monitored by oesophageal probe and maintained between 32°C and 34°C during 48 hours and followed by strictly passive rewarming. During this phase of treatment, patients will receive deep sedation associated with neuromuscular blockers. Centers participating to the trial will have expertise in cooling methods.
  Arms: Hypothermia
Procedure: local recommendations and guidelines — Investigational procedure:
  This study evaluates the impact of mild induced hypothermia (32-34°C) during 48 hours followed by passive rewarming according to recommendations described in appendix. All treatment will be according to local recommendations and guidelines of medical societies and literature. Physicians are advised to use these recommendations; however, the best treatment option for the individual patient should be used.
  Controls will receive standard care and will be also be deeply sedated for 48 hours.
  Arms: No hypothermia

SUMMARY:
Bacterial meningitis is a severe infection of the envelope which surrounds the brain. It is sometimes responsible for a cerebral oedema mattering with a loss of consciousness (coma). The usual treatment of this affection is based on the antibiotic therapy, anti-inflammatory drug and resuscitation measures in intensive care setting but the prognosis of comatose patients remains poor.

Moderate hypothermia (body temperature is downed between 32 and 34°C°) made the proof of its efficiency in certain cerebral pathologies (notably the cerebral distress after cardiac arrest or oxygen lack in neonates) but was never evaluated in meningitis. In meningitis animal studies and in severe traumatic brain injury, moderate hypothermia is able to diminish cerebral oedema and brain inflammation.

Thus, the objective of this study is to compare two strategies: only usual care or usual care completed by moderate hypothermia. The body temperature will be lowered between 32 and 34°C by means of a catheter placed in a big vein and connected to a machine in which circulates a cold liquid, or by means of an external cooling (ice-cold blanket, ice packs placed on the body). Whatever technique is chosen, the technique is perfectly mastered by the teams which take charge of the patients. After 48 hours, the technique of hypothermia will be suspended and body temperature will return passively and gradually to normal.

The investigators believe that moderate hypothermia will improve the prognosis of the most severe patients.

DETAILED DESCRIPTION:
Investigational procedure:

This study evaluates the impact of mild induced hypothermia (32-34°C) during 48 hours followed by passive rewarming according to recommendations described in appendix. All treatment will be according to local recommendations and guidelines of medical societies and literature. Physicians are advised to use these recommendations; however, the best treatment option for the individual patient should be used.

Mild Induced hypothermia:

Investigators are advised to use the cooling techniques as used in patients with cardiac arrest. Thus, the choice of cooling method will be left to investigators. Hypothermia will be induced by cold saline infusion as described in appendix 5 [6, 48]. Core temperature will be monitored by oesophageal probe and maintained between 32°C and 34°C during 48 hours and followed by strictly passive rewarming. During this phase of treatment, patients will receive deep sedation associated with neuromuscular blockers. Centers participating to the trial will have expertise in cooling methods.

Controls:

Controls will receive standard care and will be also be deeply sedated for 48 hours.

ELIGIBILITY:
INCLUSION CRITERIA:

* Subject is 18 years of age or older
* Clinically suspected community-acquired bacterial meningitis (More than 100 white blood cells in CSF and a glucose CSF/Blood ratio of 1/3 or less, or a CSF protein level above 2,2 g/L.)
* Presence of micro-organisms on CSF Gram's stain examination
* Positive soluble antigen or PCR for S. pneumoniae or N. meningitides
* Positive CSF cultures
* Score on Glasgow Coma Score < 8
* Patient received appropriate antimicrobial therapy (according to recommendations)
* If present, legally acceptable representative has provided written and dated informed consent to participate in the study.

EXCLUSION CRITERIA:

* Glasgow Coma Score < 8 for more than 12 hours
* Patients with HIV positivity: positive cryptococcal antigen in blood or CSF; Cerebral abscess
* pregnancy
* Subject has been designated as "not full support", "do not resuscitate" or equivalent status which prohibits the use of life supporting interventions thereby limiting options available
* Subject admitted for a clinical situation in which induced hypothermia is recommended
* Purpura fulminancy, defined as septic shock with extensive necrotizing purpura and disseminated intravascular coagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-03; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with unfavorable outcome (defined as score on Glasgow outcome Scale < 5) at 3 months after admission. | 3 months

SECONDARY OUTCOMES:
Mortality (assessed on day 14 after admission, day 28, total in-hospital mortality, and at 3 and 6 months) | 6 months
ICU length of stay | 6 months
Score on GOS at ICU discharge and 6 months after admission | 6 months
Neurological examination at discharge and 6 months after admission | 6 months
Neuropsychological outcome at 6 months in a subset of centres; patient will be tested with a neuropsychological test battery described previously | 6 months
MRC score on ICU discharge | 3 months
Prevalence of status EPILEPTISIS | 6 months
Prevalence of infections (aspiration pneumonia and nosocomial infections) | 6 months
Potential hypothermia related side effects as cardiac arrhythmia, electrolyte balance, hyperglycemia, bleeding, acute pancreatitis (see definitions further). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: MOURVILLIER Bruno, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Bichat Claude Bernard, Paris, France

REFERENCES:
- [Derived] Mourvillier B, Tubach F, van de Beek D, Garot D, Pichon N, Georges H, Lefevre LM, Bollaert PE, Boulain T, Luis D, Cariou A, Girardie P, Chelha R, Megarbane B, Delahaye A, Chalumeau-Lemoine L, Legriel S, Beuret P, Brivet F, Bruel C, Camou F, Chatellier D, Chillet P, Clair B, Constantin JM, Duguet A, Galliot R, Bayle F, Hyvernat H, Ouchenir K, Plantefeve G, Quenot JP, Richecoeur J, Schwebel C, Sirodot M, Esposito-Farese M, Le Tulzo Y, Wolff M. Induced hypothermia in severe bacterial meningitis: a randomized clinical trial. JAMA. 2013 Nov 27;310(20):2174-83. doi: 10.1001/jama.2013.280506. PMID 24105303